CLINICAL TRIAL: NCT00262730
Title: A Phase II Trial of Radiation Plus Temozolomide Followed by Adjuvant Temozolomide and Poly-ICLC in Patients With Newly Diagnosed Glioblastoma Multiforme
Brief Title: Radiation Therapy and Temozolomide Followed by Temozolomide and Poly ICLC in Treating Patients With Newly Diagnosed GBM
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NABTT-0501; U01CA062475 (NIH); NABTT-0501 CDR0000454915; NA_00001963 (Other: JHM IRB)
Record Dates: First submitted 2005-12-06; First posted 2005-12-07 (Estimated); Results first posted 2014-07-16 (Estimated); Last update posted 2019-06-12 (Actual); Status verified 2019-05

CONDITIONS: Glioblastoma Multiforme
Keywords: adult glioblastoma; adult giant cell glioblastoma; adult gliosarcoma
MeSH Terms: conditions — Glioblastoma; Gliosarcoma | interventions — poly ICLC; Temozolomide; Radiotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Treatment Arm (Experimental): RT + TMZ 6wks, followed by
  poly ICLC, temozolomide, radiation: radiation therapy
  Interventions: Drug: poly ICLC; Drug: temozolomide; Radiation: radiation therapy

INTERVENTIONS:
Drug: poly ICLC — 20 mcg/kg 3x each week (Maintenance cycles)
  Other Names: Holtonol
Drug: temozolomide — daily 75mg/m2 6wks concomitant therapy Wk 1 - days 1-5 150-200 mg/m2 maintenance cycles (adjuvant)
  Other Names: Temodar
Radiation: radiation therapy — RT: 60 Gy (6 weeks) concomitant therapy
  Other Names: RT

SUMMARY:
RATIONALE: Radiation therapy uses high-energy x-rays to kill tumor cells. Drugs used in chemotherapy, such as temozolomide, work in different ways to stop the growth of tumor cells, either by killing the cells or by stopping them from dividing. Biological therapies, such as poly ICLC, may stimulate the immune system in different ways and stop tumor cells from growing. Giving poly ICLC after radiation therapy and temozolomide may stop any remaining tumor cells from growing.

PURPOSE: This phase II trial is studying how well giving radiation therapy together with temozolomide followed by temozolomide and poly ICLC works in treating patients with newly diagnosed glioblastoma multiforme.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Evaluate the safety and efficacy of radiation plus low-dose temozolomide followed by adjuvant temozolomide and intramuscular poly ICLC for adult patients with newly diagnosed glioblastoma multiforme.

Secondary

* Estimate the frequency of toxicity associated with this treatment regimen.

OUTLINE: This is an open-label, multicenter study.

* Induction chemoradiotherapy: Patients undergo radiotherapy once daily, 5 days a week, for 6 weeks. During the same 6 weeks, patients also receive oral temozolomide once daily. Four weeks later, patients are evaluated for disease progression. Patients with progressive disease are removed from the study. Patients with no progressive disease proceed to maintenance therapy.
* Maintenance therapy: Patients receive oral temozolomide once daily on days 1-5 (week 1). Patients also receive poly ICLC intramuscularly three times a week in weeks 2-8. Courses repeat every 9 weeks in the absence of disease progression or unacceptable toxicity.

After completion of study therapy, patients are followed every 2 months for survival.

PROJECTED ACCRUAL: A total of 96 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed supratentorial grade IV astrocytoma (glioblastoma multiforme) by biopsy or resection within the past 3 months

PATIENT CHARACTERISTICS:

* Karnofsky performance status ≥ 60%
* Absolute neutrophil count ≥ 1500/mm^3
* Platelet count ≥ 100,000/mm^3
* Bilirubin ≤ 1.5 mg/dL
* Transaminases ≤ 4 times above the upper limits of the institutional normal
* Creatinine ≤ 1.7 mg/dL
* Not pregnant or breast-feeding
* Patients must agree to follow acceptable birth control methods to avoid conception
* Negative pregnancy test
* Patients must have a Mini Mental State Exam score of ≥ 15
* No serious concurrent infection or medical illness which would jeopardize the ability of the patient to receive the treatment outlined in this protocol with reasonable safety
* Patients with a concurrent or prior malignancy are ineligible unless they are patients with curatively treated carcinoma-in-situ or basal cell carcinoma of the skin

  * Patients who have been free of disease (any prior malignancy) for ≥ five years are eligible for this study
* Patients requiring ongoing therapy for psychoses with antipsychotic medications at the time of enrollment will be ineligible

PRIOR CONCURRENT THERAPY:

* Patients must not have received prior radiation therapy, chemotherapy, immunotherapy or therapy with biologic agent (including immunotoxins, immunoconjugates, antisense, peptide receptor antagonists, interferons, interleukins, TIL, LAK or gene therapy), or hormonal therapy for their brain tumor

  * Prior glucocorticoid therapy is allowed
* Patients must be willing to forego other cytotoxic and non-cytotoxic drug therapy against the tumor while being treated with poly ICLC plus temozolomide on this protocol
* No other concurrent therapy for their tumor (i.e., chemotherapeutics or investigational agents)
* Patients who have received prior Gliadel wafers are not eligible for this study
* No concurrent prophylactic filgrastim (G-CSF)
* No concurrent electron, particle, implant, or stereotactic radiosurgery boost

Ages: 18 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 97 (Actual)
Dates: Start 2006-01; Primary Completion 2009-08 (Actual); Study Completion 2010-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Myrna Rosenfeld, MD, PhD, Study Chair — Abramson Cancer Center at Penn Medicine
Locations (9):
- United States (9):
  - Lurleen Wallace Comprehensive Cancer at University of Alabama-Birmingham, Birmingham, Alabama
  - H. Lee Moffitt Cancer Center and Research Institute at University of South Florida, Tampa, Florida
  - Winship Cancer Institute of Emory University, Atlanta, Georgia
  - Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins, Baltimore, Maryland
  - Massachusetts General Hospital Cancer Center, Boston, Massachusetts
  - Josephine Ford Cancer Center at Henry Ford Hospital, Detroit, Michigan
  - Wake Forest University Comprehensive Cancer Center, Winston-Salem, North Carolina
  - Cleveland Clinic Taussig Cancer Center, Cleveland, Ohio
  - Abramson Cancer Center of the University of Pennsylvania, Philadelphia, Pennsylvania

REFERENCES:
- [Result] Rosenfeld MR, Chamberlain MC, Grossman SA, Peereboom DM, Lesser GJ, Batchelor TT, Desideri S, Salazar AM, Ye X. A multi-institution phase II study of poly-ICLC and radiotherapy with concurrent and adjuvant temozolomide in adults with newly diagnosed glioblastoma. Neuro Oncol. 2010 Oct;12(10):1071-7. doi: 10.1093/neuonc/noq071. Epub 2010 Jul 8. PMID 20615924

RESULTS

PARTICIPANT FLOW:
Recruitment Details: outpatient clinic
Groups:
- Treatment Arm - All Subjects: poly ICLC, temozolomide, radiation: radiation therapy
  poly ICLC : 20 mcg/kg 3x each week (Maintenance cycles)
  temozolomide : daily 75mg/m2 6wks concomitant therapy Wk 1 - days 1-5 150-200 mg/m2 maintenance cycles (adjuvant)
  radiation therapy : RT: 60 Gy (6 weeks) concomitant therapy
Period: Overall Study
Arm/Group | Treatment Arm - All Subjects
Started | 97
Completed | 97
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Treatment Arm - All Subjects
Number analyzed (Participants) | 97
Age, Continuous [Median (Full Range); unit: years] | 56.6 [21 to 85]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 37
  Male | 60
Karnofsky Performance Status [Number; unit: Units on a scale] — 100 normal no complaints no disease 90 capable of normal activity few symptoms/disease 80 normal activity with some difficulty some symptoms or signs 70 caring for self not capable of normal activity or work 60 requiring some help can take care of most personal requirements 50 requires help often requires frequent medical care 40 disabled requires special care and help 30 severely disabled hospital admission indicated but no risk of death 20 very ill urgently requiring admission requires supportive measures or treatment 10 moribund rapidly progressive fatal disease processes 0 death
  Units on a scale
    100 | 34
    90 | 45
    80 | 12
    70 | 3
    60 | 3
Extent of surgery [Number; unit: Patient]
  Biopsy | 18
  Craniotomy | 79
time from diagnosis to radiotherapy [Median (Full Range); unit: weeks] | 4.4 [2 to 12.6]
Baseline Mini-Mental State Examiniation (MMSE) Score [Number; unit: Scores on a Scale] — The mini-mental state examination (MMSE) is a 30-point questionnaire test used to screen for cognitive impairment. Commonly used to screen for dementia. It is also used to estimate the severity of cognitive impairment and to follow the course of cognitive changes in an individual over time. The MMSE test includes simple questions and problems in a number of areas: the time and place of the test, repeating lists of words, arithmetic such as the serial sevens, language use and comprehension, and basic motor skills. The Higher your score, the higher your function.
  Scores on a Scale
    30 | 56
    27-29 | 30
    Less than or equal 26 | 11
Corticosteroid Therapy [Number; unit: Participant]
  Yes | 70
  No | 26
  Missing Data | 1
Histologic Diagnosis [Number; unit: Patient]
  Glioblastoma | 94
  Anaplastic Astrocytoma | 1
  Other | 2

OUTCOME MEASURES:

1. Primary Outcome: Survival
Description: survival time is defined from time of histological diagnosis to death occurrence.
Time Frame: 30 months
Population: all patients who were treated were analyzed (intent to treat)
Measure: Mean (95% Confidence Interval); unit: months
Arm/Group | Treatment Arm - All Subjects
Number analyzed (Participants) | 97
months | 17.2 [15.4 to 19.3]
Statistical Analysis 1: Comparison: Treatment Arm - All Subjects; Test type: Non-Inferiority or Equivalence — study design has 85% power to detect 25% deduction in hazard rate compared to EORTC Phase 3 results; p > .1, Log Rank; Hazard Ratio (HR) = 0.8, 95% CI 2-sided [0.8 to 0.85], Standard Deviation .025

ADVERSE EVENTS:
Time Frame: While on Treatment
Groups:
- Treatment Arm All Subjects: poly ICLC, TMZ, RT: poly ICLC : 20 mcg/kg 3x each week (Maintenance cycles) TMX : daily 75mg/m2 6wks concomitant therapy Wk 1 - days 1-5 150-200 mg/m2 maintenance cycles (adjuvant) RT : RT: 60 Gy (6 weeks) concomitant therapy
  AEs Grades 4 with Attributions of Possible, probably or definitely related to TMZ AND poly-ICLI
Arm/Group | Treatment Arm All Subjects
Serious Adverse Events (participants affected / at risk) | 20/97
Other Adverse Events (participants affected / at risk) | 97/97
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment Arm All Subjects (N=97)
Diarrhea (Gastrointestinal disorders) | 1 (1)
fatigue (General disorders) | 3 (3)
muscle weakness, generalized (Musculoskeletal and connective tissue disorders) | 1 (1)
nausea (Nervous system disorders) | 1 (1)
vomiting (Gastrointestinal disorders) | 1 (1)
rash (Skin and subcutaneous tissue disorders) | 2 (2) — desquamation
aspartate aminotransferase increased (Investigations) | 1 (1)
febrile neutropenia (Blood and lymphatic system disorders) | 2 (2)
hemoglobin increased (Blood and lymphatic system disorders) | 2 (2)
Lung infection (Infections and infestations) | 1 (1) — pneumonia
leukopenia (Blood and lymphatic system disorders) | 16 (16)
Neutrophils/granulocytes (ANC/AGC) (Investigations) | 20 (20)
platelet count decreased (Investigations) | 9 (9)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment Arm All Subjects (N=97)
Alkaline phosphatase increased (Investigations) | 19 (66)
allergic reaction (Immune system disorders) | 2 (2)
allergic rhinitis (Respiratory, thoracic and mediastinal disorders) | 4 (4)
anorexia (Metabolism and nutrition disorders) | 28 (35)
arthritis (Musculoskeletal and connective tissue disorders) | 1 (1)
ascites (Gastrointestinal disorders) | 1 (1)
ataxia (Nervous system disorders) | 10 (12)
ear and labyrinth disorder (Ear and labyrinth disorders) | 4 (4) — other
blood bicarbonate decreased (Investigations) | 10 (13)
bruising (Injury, poisoning and procedural complications) | 12 (17)
ischemia cerebrovascular (Nervous system disorders) | 3 (3)
cataract (Eye disorders) | 1 (1)
cognitive disturbance (Nervous system disorders) | 2 (2)
colitis (Gastrointestinal disorders) | 3 (3)
confusion (Nervous system disorders) | 18 (26)
constipation (Gastrointestinal disorders) | 38 (52)
cough (General disorders) | 18 (22)
creatinine increased (Investigations) | 3 (3)
cushingoid (Endocrine disorders) | 8 (8)
cystitis (Renal and urinary disorders) | 1 (1)
dehydration (Metabolism and nutrition disorders) | 3 (3)
periodontal disease (Gastrointestinal disorders) | 1 (1)
dermatology/skin (Skin and subcutaneous tissue disorders) | 5 (5)
diarrhea (Gastrointestinal disorders) | 13 (19)
distension/bloating (Gastrointestinal disorders) | 1 (1)
dizziness (Nervous system disorders) | 24 (28)
dry eye (Eye disorders) | 3 (3)
dry mouth (Gastrointestinal disorders) | 2 (2)
dry skin (Skin and subcutaneous tissue disorders) | 4 (5)
dysphagia (Gastrointestinal disorders) | 3 (3)
dyspnea (Respiratory, thoracic and mediastinal disorders) | 15 (18)
edema (General disorders) | 5 (5) — head and neck
edema (General disorders) | 19 (28) — limbs
encephalopathy (Nervous system disorders) | 1 (1)
endocrine (Endocrine disorders) | 1 (1)
extremity - lower (gait/walking) (Musculoskeletal and connective tissue disorders) | 1 (1) — gait disturbance
fatigue (General disorders) | 70 (112)
febrile neutropenia (Blood and lymphatic system disorders) | 3 (3)
fever (General disorders) | 9 (13) — in absence of neutropenia
flu like symptoms (General disorders) | 3 (4)
flushing (Vascular disorders) | 1 (1)
fracture (Injury, poisoning and procedural complications) | 1 (1)
gastritis (Gastrointestinal disorders) | 3 (3)
gastrointestinal (Gastrointestinal disorders) | 4 (8)
hyperglycemia (Metabolism and nutrition disorders) | 1 (3)
anemia (Blood and lymphatic system disorders) | 71 (760)
alopecia (Skin and subcutaneous tissue disorders) | 39 (39)
hearing (Ear and labyrinth disorders) | 4 (4) — w/o baseline audiogram & no monitoring program
dyspepsia (Gastrointestinal disorders) | 12 (12)
hemoglobin increase (Blood and lymphatic system disorders) | 2 (2)
hemorrhage (Nervous system disorders) | 1 (1) — CNS
esophageal hemorrhage (Infections and infestations) | 1 (1)
rectal hemorrhage (Gastrointestinal disorders) | 1 (1)
hemorrhage (Renal and urinary disorders) | 1 (1) — urinary
hemorrhage (Respiratory, thoracic and mediastinal disorders) | 2 (2) — nose
hiccups (Respiratory, thoracic and mediastinal disorders) | 1 (1)
hot flashes (Vascular disorders) | 2 (2)
hydrocephalus (Nervous system disorders) | 4 (4)
hypercalcemia (Metabolism and nutrition disorders) | 6 (9)
hyperglycemia (Metabolism and nutrition disorders) | 65 (246)
hyperkalemia (Metabolism and nutrition disorders) | 15 (32)
hypermagnesemia (Metabolism and nutrition disorders) | 18 (27)
hypernatremia (Metabolism and nutrition disorders) | 12 (20)
hyperpigmentation (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
hypertension (Vascular disorders) | 2 (2)
hypocalcemia (Metabolism and nutrition disorders) | 18 (33)
hypoglycemia (Metabolism and nutrition disorders) | 20 (41)
hypokalemia (Metabolism and nutrition disorders) | 18 (32)
hypomagnesemia (Metabolism and nutrition disorders) | 6 (9)
hyponatremia (Metabolism and nutrition disorders) | 20 (53)
hypotension (Vascular disorders) | 7 (9)
hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 (1)
International Normalized Ratio of prothrombin time (Hepatobiliary disorders) | 2 (2)
urinary incontinence (Renal and urinary disorders) | 4 (5)
infection (Infections and infestations) | 42 (45) — bladder (urinary)
insomnia (Psychiatric disorders) | 20 (26)
injury (Injury, poisoning and procedural complications) | 1 (1) — intra-operative brain injury
joint function (Musculoskeletal and connective tissue disorders) | 2 (2)
leukocytes (Blood and lymphatic system disorders) | 2 (2) — total white blood cell count
libido decreased (Psychiatric disorders) | 2 (2)
lumbar spine range of motion decreased (Musculoskeletal and connective tissue disorders) | 1 (1)
memory impairment (Nervous system disorders) | 27 (32)
mood alteration (Psychiatric disorders) | 36 (39)
mucositis oral (Gastrointestinal disorders) | 11 (12)
muscle weakness, generalized or specific area (Musculoskeletal and connective tissue disorders) | 33 (43)
soft tissue (Musculoskeletal and connective tissue disorders) | 5 (7)
nail changes (Skin and subcutaneous tissue disorders) | 1 (1)
paranasal sinus reaction (Respiratory, thoracic and mediastinal disorders) | 2 (2)
nausea (Gastrointestinal disorders) | 41 (64)
neurological disorder (Nervous system disorders) | 8 (8)
neuropathy (Nervous system disorders) | 58 (80)
Neutrophils/granulocytes (ANC/AGC) (Investigations) | 3 (3)
obstruction (Renal and urinary disorders) | 2 (2) — ureter, bladder
ocular/vision disorder (Eye disorders) | 2 (2)
diplopia (double vision) (Eye disorders) | 3 (4)
lymphopenia (Blood and lymphatic system disorders) | 1 (1)
otitis (Ear and labyrinth disorders) | 2 (2) — external ear, middle ear
PLTS (Blood and lymphatic system disorders) | 59 (468)
PO4 (Blood and lymphatic system disorders) | 19 (31)
PTT (Investigations) | 4 (10)
pain - abdomen (Gastrointestinal disorders) | 2 (2)
pain - back (Musculoskeletal and connective tissue disorders) | 8 (10)
pain - bone (Musculoskeletal and connective tissue disorders) | 1 (1)
pain - breast (Reproductive system and breast disorders) | 1 (1)
pain - cardiac/heart/chest (Cardiac disorders) | 3 (3)
pain - chest/thorax (General disorders) | 4 (6)
pain - dental/teeth/peridontal (Gastrointestinal disorders) | 1 (1)
pain - external ear (Ear and labyrinth disorders) | 1 (1)
pain - extremity (Musculoskeletal and connective tissue disorders) | 14 (16)
pain - eye (Eye disorders) | 2 (2)
headache (Nervous system disorders) | 51 (80)
pain - joint (Musculoskeletal and connective tissue disorders) | 16 (21)
pain - middle ear (Ear and labyrinth disorders) | 3 (3)
pain - muscle (Musculoskeletal and connective tissue disorders) | 17 (23)
pain - neck (Musculoskeletal and connective tissue disorders) | 6 (6)
pain - oral (Gastrointestinal disorders) | 1 (1)
pain - other (General disorders) | 4 (4)
pain - scalp (Skin and subcutaneous tissue disorders) | 3 (3)
pain - skin (Skin and subcutaneous tissue disorders) | 3 (3)
pain - stomach (Gastrointestinal disorders) | 2 (2)
palpitations (Cardiac disorders) | 4 (4)
personality/behavioral disorder (Psychiatric disorders) | 1 (1)
photosensitivity (Eye disorders) | 1 (1)
platelets (Blood and lymphatic system disorders) | 2 (3)
pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1 (1)
hyperkalemia (Metabolism and nutrition disorders) | 1 (1)
hypokalemia (Metabolism and nutrition disorders) | 3 (4)
pruritus/itching (Skin and subcutaneous tissue disorders) | 9 (11)
psychosis (Psychiatric disorders) | 3 (3)
pulmonary/upper respiratory (Respiratory, thoracic and mediastinal disorders) | 2 (2)
pyramidal tract dysfunction (Nervous system disorders) | 1 (1)
purpura (Skin and subcutaneous tissue disorders) | 2 (3)
rash - acneiform (Skin and subcutaneous tissue disorders) | 4 (4)
rash (Injury, poisoning and procedural complications) | 20 (20) — associated with radiation (chemoradiation & radiation)
rash - desquamation (Skin and subcutaneous tissue disorders) | 20 (27)
rigors/chills (General disorders) | 5 (7)
SGOT/AST (Investigations) | 18 (37)
SGPT/ALT (Investigations) | 34 (131)
seizure (Nervous system disorders) | 34 (68)
skin breakdown/decubitus ulcer (Skin and subcutaneous tissue disorders) | 1 (1)
hyponatremia (Metabolism and nutrition disorders) | 2 (2)
somnolence (Nervous system disorders) | 4 (4)
speech impairment (Nervous system disorders) | 22 (34) — dysphasia or aphasia
supraventricular and nodal arrhythmia (Cardiac disorders) | 1 (1) — atrial fibrillation
supraventricular and nodal arrhythmia (Cardiac disorders) | 1 (1) — atrial tachycardia/paroxysmal atrial tachycardia
supraventricular and nodal arrhythmia (Cardiac disorders) | 1 (1) — sinus tachycardia
sweating (diaphoresis) (Skin and subcutaneous tissue disorders) | 3 (3)
syncope (Nervous system disorders) | 3 (3)
syndromes - other (General disorders) | 1 (1)
taste alteration (Gastrointestinal disorders) | 11 (12) — dysgeusia
thrombosis/thrombus/embolism (Nervous system disorders) | 12 (14)
tinnitus (Ear and labyrinth disorders) | 7 (9)
total bilirubin (Investigations) | 3 (5)
tremor (Nervous system disorders) | 6 (6)
ulceration (Gastrointestinal disorders) | 1 (2)
uric acid (Metabolism and nutrition disorders) | 6 (13)
urinary frequency (Renal and urinary disorders) | 3 (3)
urinary retention (Renal and urinary disorders) | 3 (3)
urticaria (Skin and subcutaneous tissue disorders) | 1 (1)
vaginal discharge (Reproductive system and breast disorders) | 1 (1)
vascular - other (Vascular disorders) | 2 (3)
vision - blurred (Eye disorders) | 16 (20)
vision - flashing lights/floaters (Eye disorders) | 4 (4)
voice changes (Respiratory, thoracic and mediastinal disorders) | 2 (2) — hoarseness, loss or alteration in voice, laryngitis
white blood cells (Investigations) | 64 (793)
watery eye (Eye disorders) | 1 (1) — epiphora, tearing
weight gain (Metabolism and nutrition disorders) | 2 (2)
weight loss (Metabolism and nutrition disorders) | 10 (10)

LIMITATIONS AND CAVEATS:
"Other Adverse Events" not reported for this study. Only serious(grade 3/4)related to either TMZ and/or Poly were reported. Subjects may have experienced grade 1 and grade 2 other adverse event but they have no bearing on clinical outcome of agent

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No